CLINICAL TRIAL: NCT04307914
Title: Focused Ultrasound and RadioTHERapy for Noninvasive Palliative Pain Treatment in Patients With Bone Metastases
Acronym: FURTHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Turku University Hospital (Other Government); Universitätsklinikum Köln (Other); University of Roma La Sapienza (Other); Istituto Ortopedico Rizzoli (Other); University of Bologna (Other); Isala (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL71303.041.19
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Bone Metastases; Bone Neoplasm; Bone Lesion; Bone Cancer; Pain; Cancer Induced Bone Pain; Quality of Life; Tumor; Neoplasm Metastasis
Keywords: Bone Metastases; Cancer Induced Bone Pain; Pain palliation; Raiotherapy; Radiation oncology; Noninvasive; MR-HIFU; MRgFUS; HIFU; Focused Ultrasound
MeSH Terms: conditions — Bone Neoplasms; Pain; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A total of 216 patients with painful bone metastases will be randomized in a 1:1:1 ratio to receive EBRT only, MR-HIFU only, or EBRT followed by MR-HIFU. In addition, data of around 60-90 patients will be captured within the FURTHER Registry arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- External Beam Radiotherapy (Active Comparator): In the control arm, patients will undergo standard radiotherapy for painful bone metastases.The radiation schedule is at the discretion of the treating radiation oncologist.
  Interventions: Radiation: External beam radiotherapy
- MR-HIFU (Experimental): In the intervention arm, patients will be offered MR-HIFU treatment instead of standard radiotherapy. Treatment will be given following the international guidelines for MR-HIFU.
  Interventions: Procedure: MR-HIFU
- Combination EBRT + MR-HIFU (Experimental): In the combination arm, patients will undergo standard radiotherapy followed by MR-HIFU in a short timeframe.
  Interventions: Radiation: External beam radiotherapy; Procedure: MR-HIFU

INTERVENTIONS:
Radiation: External beam radiotherapy — The current standard of care for patients with uncomplicated painful bone metastases is palliative locoregional external beam radiotherapy, often in combination with systemic therapy and analgesics.
  Arms: Combination EBRT + MR-HIFU; External Beam Radiotherapy
Procedure: MR-HIFU — MR-HIFU is a non-invasive treatment modality that delivers acoustic energy to heat tissue to ablative temperatures of more than 60°C. The combination of focused ultrasound with magnetic resonance imaging (MRI) enables physicians to perform localized tumor tissue ablation, with real-time temperature monitoring using magnetic resonance (MR) thermometry.
  Other Names: MRgFUS; MR guided High Intensity Focused Ultrasound
  Arms: Combination EBRT + MR-HIFU; MR-HIFU

SUMMARY:
The FURTHER study aims to evaluate the effectiveness and cost-effectiveness of MR-HIFU (alone or in combination with EBRT) compared to EBRT alone, the standard-of-care, as a palliative treatment option to relieve CIBP. The FURTHER study consists of a multicenter, three-armed randomized controlled trial (FURTHER RCT) and a patient registry arm (FURTHER Registry), which will be performed in six hospitals in four European countries.

DETAILED DESCRIPTION:
Rationale: Cancer induced bone pain (CIBP) as a result of bone metastases strongly interferes with quality of life and daily functioning of patients with advanced cancer. The current standard of care for patients with painful bone metastasis includes palliative external beam radiotherapy (EBRT). While EBRT is a well-established treatment option, it takes up to 4-6 weeks for EBRT to induce optimal pain relief, and 30-40% of patients do not respond to EBRT. Pain palliation may be improved by including magnetic resonance image guided high intensity focused ultrasound (MR-HIFU) as alternative or in addition to EBRT.

Objective: The FURTHER study aims to evaluate the effectiveness and cost-effectiveness of MR-HIFU (alone or in combination with EBRT), as a palliative treatment option to relieve CIBP.

Study design: The FURTHER study consists of a prospective, multicenter, three-armed randomized controlled trial (FURTHER RCT) and a patient registry arm (FURTHER Registry), performed in six hospitals in four European countries, all of which are partners in the FURTHER consortium. The UMC Utrecht is coordinating center. Within the FURTHER RCT, a total of 216 patients with painful bone metastases will be included. These patients will be randomized in a 1:1:1 ratio to receive EBRT only, MR-HIFU only, or EBRT followed by MR-HIFU. In the Netherlands, we expect to enroll a minimum of 70 patients, and a maximum of 120 patients in three Dutch study sites. Within the FURTHER Registry, data of around 60-90 patients will be captured.

Study population: The study will be performed in male and female adult (≥ 18 years) cancer patients capable of giving informed consent having painful non-spinal bone metastases (pain score on Numerical Rating Scale (NRS) ≥ 4).

Intervention: The intervention under study is MR-HIFU alone or in combination with EBRT. The intervention is aimed at rapid and persistent relief of CIBP. In the FURTHER RCT, the intervention will be compared to standard treatment EBRT.

Main study endpoints: Primary outcome of the study will be pain response at 14 days after the first day of treatment. Secondary outcomes include pain response at 14 days after inclusion, and pain scores, toxicity, adverse events, quality of life and survival in the first 6 months after treatment, and cost-effectiveness of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving informed consent
* Age ≥ 18 years
* Painful metastatic bone lesion (NRS > 2)
* Patient-localised pain with a distinct pathological substrate on recent CT/MRI
* Target lesion location is sufficiently accessible for MR-HIFU to expect clinical response, as judged by the (intervention) radiologist
* Participant has a reasonable performance score (KPS ≥ 50% or Zubrod/ECOG/WHO < 3)
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Participant is not able to fit in the MR gantry
* Need for surgery of targeted location due to (impending) pathological fracture
* Unavoidable critical structures or dense tissues in target area
* Contra-indications for MRI or sedation/anesthesia
* Clinically relevant medical history or physical findings that could interfere with the patient's safety as judged by the treating physician
* Participant enrolled in another clinical interventional study related to bone metastases treatment or pain relief treatment

All patients meeting the FURTHER in- and exclusion criteria as described above will be included in this study, either in the FURTHER RCT or FUTHER Registry. The following inclusion criteria are used to decide upon the arm patients will participate in. If patients meet all of the following RCT inclusion criteria, they will be asked to participate in the FURTHER RCT. Alternatively, patients who do not meet one or more of these criteria will be asked to participate in the FURTHER Registry.

* Painful bone lesion (NRS ≥ 4)
* Indication for EBRT treatment of a bone lesion
* Exclusively palliative intention of EBRT treatment plan
* No previous surgery on the target location
* No neurological symptoms due to nerve involvement of target lesion
* No (impending) pathological fracture)
* EBRT replacable by MR-HIFU based on medical history or phyiscal findings judged by multidisciplinary team
* Target lesion location is completely accessible for MR-HIFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain response - 14 days after completion of treatment | 14 days
  Patient reported pain response will be based on a Numeric Rating Scale (from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable) and the pain severity index calculated from the Brief Pain Inventory (BPI) questionnaire [Cleeland 1994]. In addition, analgesic and anti-neuropathic drug use is recorded, and all opioid analgesics are expressed as the oral equivalent daily morphine use (OMED). The primary endpoint of the RCT will follow the International Consensus on Palliative Radiotherapy Endpoints for Future Clinical Trials in Bone metastases (Chow 2012). Patients will be categorized as responders when a complete or partial pain response is achieved. All other patients will be categorized as non-responders.

SECONDARY OUTCOMES:
Pain response - 14 days after inclusion | 14 days
  Patient reported pain response will be based on a Numeric Rating Scale (from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable) and the pain severity index calculated from the Brief Pain Inventory (BPI) questionnaire [Cleeland 1994]. In addition, analgesic and anti-neuropathic drug use is recorded, and all opioid analgesics are expressed as the oral equivalent daily morphine use (OMED). This endpoint will follow the International Consensus on Palliative Radiotherapy Endpoints for Future Clinical Trials in Bone metastases (Chow 2012). Patients will be categorized as responders when a complete or partial pain response is achieved. All other patients will be categorized as non-responders.
Patient reported pain scores - patient pain diary | 21 days
  Patient reported pain scores will be based on a Numeric Rating Scale (from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable). This will be assessed using a daily patient pain diary during the first 21 days after completion of treatment.
Patient reported pain scores - BPI | on baseline, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  Patient reported pain scores will be based on a Numeric Rating Scale (from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable). This will be assessed using the Brief Pain Inventory (BPI) questionnaire at 7 time points during the total follow up of 6 months.
Physician reported toxicity - CTCAE 5.0 | at 3 days, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  Assessed in seven telephone calls during the first six months following completion of treatment according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Patient reported quality of life - EORTC BM22 | on baseline, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  During the follow up time of 6 months, patients will receive the EORTC BM22 quality of life questionnaire at baseline, one, two, four and six weeks, and three and six months following completion of treatment.
Patient reported quality of life - EORTC C15-PAL | on baseline, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  During the follow up time of 6 months, patients will receive the EORTC C15-PAL quality of life questionnaire at baseline, one, two, four and six weeks, and three and six months following completion of treatment.
Patient reported quality of life - EQ-5D-5L | on baseline, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  During the follow up time of 6 months, patients will receive the EQ-5D-5L quality of life questionnaire at baseline, one, two, four and six weeks, and three and six months following completion of treatment.
Patient reported quality of life - PGIC | at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  During the follow up time of 6 months, patients will receive the Patient Global Impression of Change scale (a 7 point likert scale about overall improvement after treatment) at one, two, four and six weeks, and three and six months following completion of treatment.
Patient reported quality of life - HADS | on baseline, at 1, 2, 4 and 6 weeks, and at 3 and 6 months
  During the follow up time of 6 months, patients will receive the Hospital Anxiety and Depression Scale (HADS) questionnaire at one, two, four and six weeks, and three and six months following completion of treatment.
  Assessed among patients, patients' partners and caregivers by the Hospital Anxiety and Depression Scale (HADS) at baseline, two and four weeks, and three and six months fol-lowing completion of treatment.
Local tumour control | 3 and 6 months
  Assessed using CT and/or MRI imaging at patient discretion at three and/or six months after completion of treatment.
Cost-effectiveness of the treatment | 6 months
  A hypothetical diagnosis related group (DRG) will be calculated from the perspective of the statutory health insurance (SHI).

CONTACTS AND LOCATIONS:
Locations (6):
- TUCH Turku, Turku, Finland
- University Hospital Cologne, Cologne, Germany
- Italy (2):
  - IOR, Bologna
  - CSSP, Roma
- Netherlands (2):
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken Zwolle, Zwolle

REFERENCES:
- [Derived] Slotman DJ, Bartels MMTJ, Ferrer CJ, Bos C, Bartels LW, Boomsma MF, Phernambucq ECJ, Nijholt IM, Morganti AG, Siepe G, Buwenge M, Grull H, Bratke G, Yeo SY, Blanco Sequeiros R, Minn H, Huhtala M, Napoli A, De Felice F, Catalano C, Bazzocchi A, Gasperini C, Campanacci L, Simoes Correa Galendi J, Muller D, Braat MNGJA, Moonen C, Verkooijen HM; FURTHER consortium. Focused Ultrasound and RadioTHERapy for non-invasive palliative pain treatment in patients with bone metastasis: a study protocol for the three armed randomized controlled FURTHER trial. Trials. 2022 Dec 29;23(1):1061. doi: 10.1186/s13063-022-06942-1. PMID 36582001